CLINICAL TRIAL: NCT02534194
Title: Gestational Age Assessment Tool for Newborn Babies
Brief Title: Gestational Age Assessment Tool
Acronym: GestATion
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 15020
Record Dates: First submitted 2015-08-04; First posted 2015-08-27 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Immature Newborn; Premature Birth
Keywords: Gestation; Premature; Infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newborn Infant: Newborn babies (within 7 days of birth) born between 23-42 weeks.
  Interventions: Other: Image acquisition

INTERVENTIONS:
Other: Image acquisition — Images of baby's face (including ear) and feet

SUMMARY:
In the UK and worldwide many babies are born without carers knowing their gestation as the mothers will not have had good antenatal care. It is possible to estimate gestation but this requires a detailed clinical exam. The investigators wish to improve this by using software analysis to pick out features of the baby (face and foot) to try and estimate the gestation of the baby once it is born. The investigators will also look explore if the software can distinguish the normal face or a baby in discomfort.

Good estimation of gestation can result in more targeted management of the baby. The investigators will capture the images of newborn babies, from a variety of gestations, and use this dataset to teach the software to estimate gestational age and level of discomfort.

DETAILED DESCRIPTION:
Clinical techniques for the calculation of gestation include fetal ultrasound and clinical assessment tools, such as the Ballard Score, following birth. These techniques are rarely available (ultrasound which is expensive and requires trained users) or require significant training (Ballard) which makes them unsuitable for large scale assessment in many low-middle income (LMI) countries. In the UK, the gestational age of babies of mothers with no antenatal care requires a detailed clinical examination which can lack accuracy. Clinical assessment of postnatal gestational age utilises anatomical characteristics of the face, ear and foot during newborn development. There is an element of subjectiveness which reduces the precision of such an assessment which is only reduced with significant training and experience. Simpler techniques of postnatal gestational age assessment such as anthropometric measures are time consuming and lack the accuracy required. Emerging evidence suggests that gestational age can be calculated postnatally by measuring the newborn foot length and comparing to population appropriate charts. However, when used on their own, the specificity and sensitivity are still below acceptable limits to allow universal adoption.

New software-based analytical techniques now make it possible to perform fully automatic recognition of facial actions and dimensions. The investigators have developed techniques that allow live video facial feature identification and measurement using advanced analytical techniques of muscle actions. These techniques have been used for facial expression analysis as well as automated facial feature localization. The investigators propose that the same analysis could be used to create a unique gestational age assessment tool using a simple brief video clip of the newborns' face and foot.

Accurate assessment of gestational age, especially in LMI countries, could ensure high risk newborns receive appropriate low cost interventions to reduce morbidity and mortality. In the UK this could allow better estimation of babies born to mothers with no antenatal care where the gestational age is unclear. We propose a smartphone based, ethnic appropriate, combined face and foot video analysis tool to accurately determine gestational age of the newborn. Such a system could adapted to incorporate pain assessment tools to help inform treatment options and study new therapies.

ELIGIBILITY:
Inclusion Criteria:

* Where the baby's gestational age is known (based on antenatal care)
* With written informed parental consent.

Exclusion Criteria:

* No parental consent
* Babies undergoing palliative care

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn babies within 7 days of birth recruited from Nottingham University Hospitals NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-08; Primary Completion 2018-04-15 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Software analysis tool estimates the gestational age of a newborn baby to within 1 week of its actual gestation | 12 months

SECONDARY OUTCOMES:
Quantification of pain from facial features during uncomfortable procedures. | 12 months
  Comparison with two pain scores, the neonatal Pain Assessment Tool (PAT, scored 0 (no pain) to 10 (significant pain)) and the Neonatal Infant Pain Scale (NIPS, scored 0 (no pain) to 7 (significant pain)). The software will be calibrated from these pain scores. This approach hasn't previously been performed so the software scoring system will be developed alongside these commonly used measures.

CONTACTS AND LOCATIONS:
Overall Officials: Don Sharkey, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom